CLINICAL TRIAL: NCT00629213
Title: Metabolic Syndrome and Its Single Traits as Risk Factors of Diabetes in People With Impaired Glucose Tolerance: The STOP-NIDDM Trial
Brief Title: Metabolic Syndrome Risk Factor in IGT: STOP-NIDDM Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GWT-TUD GmbH (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: Canadian: ACRI02; Bay g 5421
Record Dates: First submitted 2008-02-22; First posted 2008-03-05 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2008-03

CONDITIONS: Metabolic Syndrome
Keywords: prevention,; type 2 diabetes,; metabolic syndrome,; acarbose treatment
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus, Type 2 | interventions — Acarbose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: acarbose
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: acarbose
  Arms: 1
Drug: placebo
  Arms: 2

SUMMARY:
The aim of the study was to analyse the independent and joint effects of the components of the metabolic syndrome (MetS) on the incidence of diabetes in people with impaired glucose tolerance (IGT) and to assess the effect of acarbose by MetS status.

Double-blind placebo controlled trial, 1,368 patients, follow-up time 3.3 years. MetS by ATP III definition with fasting plasma glucose of ≥ 6.1 mmol/l as limit for impaired fasting glucose (IFG).

ELIGIBILITY:
Inclusion Criteria:

* High risk population
* Age 40 to 70 yrs.
* BMI > 25 and < 40; FPG >5.5 mmol/l and < 7.8 mmol/l; IGT in OGGT

Exclusion Criteria:

* Known type 2 diabetes
* Drug intake affecting glucose tolerance
* Any cardiovascular events within the last 6 months

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1429

PRIMARY OUTCOMES:
Incidence of newly diagnosed type 2 diabetes

SECONDARY OUTCOMES:
newly diagnosed hypertension

CONTACTS AND LOCATIONS:
Locations (1):
- GWT-TUD GmbH, Dresden, Saxony, Germany

REFERENCES:
- [Background] Chiasson JL, Josse RG, Gomis R, Hanefeld M, Karasik A, Laakso M; STOP-NIDDM Trail Research Group. Acarbose for prevention of type 2 diabetes mellitus: the STOP-NIDDM randomised trial. Lancet. 2002 Jun 15;359(9323):2072-7. doi: 10.1016/S0140-6736(02)08905-5. PMID 12086760
- [Derived] Hanefeld M, Karasik A, Koehler C, Westermeier T, Chiasson JL. Metabolic syndrome and its single traits as risk factors for diabetes in people with impaired glucose tolerance: the STOP-NIDDM trial. Diab Vasc Dis Res. 2009 Jan;6(1):32-7. doi: 10.3132/dvdr.2009.006. PMID 19156626